CLINICAL TRIAL: NCT01530737
Title: Antithrombin Enhancement May Improve Anticoagulation Efficiency in Infants Undergoing Cardiopulmonary Bypass for Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000020202
Record Dates: First submitted 2012-01-30; First posted 2012-02-10 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Cardiopulmonary Bypass
Keywords: pediatric; Antithrombin; anticoagulation efficiency; cardiac surgery
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator)
  Interventions: Other: Saline Placebo
- Active Antithrombin Group (Experimental)
  Interventions: Drug: Antithrombin III

INTERVENTIONS:
Drug: Antithrombin III — Patients randomized to receive Antithrombin concentrate will receive a dose of AT to achieve a target value of 1.2U/ml.
  Arms: Active Antithrombin Group
Other: Saline Placebo — Patients randomized to the control group will receive a placebo consisting of normal saline in a volume equivalent to the volume of antithrombin the same patient in the treatment group would have received and administered by anesthesia and perfusion in the exact same manner as the AT is administered in the treatment group.
  Arms: Control Group

SUMMARY:
The primary objective of this study is:

1. To evaluate the use of Antithrombin (AT) concentrate in infants less than one year of age undergoing cardiopulmonary bypass (CPB) for cardiac surgery

The secondary objectives of this study are:

1. To determine if the administration of AT concentrate prior to heparinization will decrease the amount of heparin required to achieve optimal anticoagulation (as defined by anti-Xa levels) during CPB
2. To determine if a decrease in activation and consumption of coagulation proteins, platelets and subsequent fibrinolysis will result in improved haemostasis following CPB
3. To determine if there will be a reduction in postoperative bleeding and associated clinical complications

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients < 1 year old with cardiac defect (acquired or congenital) requiring cardiac surgery
2. Planned cardiac surgery with cardiopulmonary bypass
3. Weight > 2.5kg at the time of surgery
4. Enrolment in the CATCH main study (REB#1000020203)

Exclusion Criteria:

1. Preoperative antithrombin activity > 85%
2. Prematurity < 36 weeks gestational age at birth
3. Preoperative use of systemic anticoagulant (i.e. heparin or warfarin at a therapeutic dose) for > 24 hours or at any time within the 48 hours prior to surgery
4. Any form of coagulopathy or thrombophilic disorder
5. Renal (blood creatinine - estimated GRF < 60ml/min/1.73m2) or clinical liver failure
6. Antithrombin replacement therapy prior to surgery
7. Repeat surgery (including previous ECMO/VAD support as prior surgery)
8. Patients refusal to provide open consent for re-use of study data

Max Age: 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Chest tube volume loss | 24 hrs post surgery
  Chest tube volume loss (mls/kg) at 24 hours in CCCU

SECONDARY OUTCOMES:
Heparin dose required to achieve target Activated Clotting Time required to go on Cardiopulmonary Bypass | 1hr prior to induction of anaestheisa (pre-surgery)
  Clinical Outcome Measure
Blood product transfusions intra-operatively and for the first 24 hours following surgery | 24hours post surgery
Clinical outcomes | 30 days post-surgery
  (inotropic support, ventilation, CCU stay, hospital stay, thrombosis)
Intraoperative coagulation profile | 5 hours after start of surgery
  (anti-Xa, heparin concentration, activated clotting time, CBC, antithrombin)
Post-operative markers of platelet activation | 24 and 72 hrs post surgery
  Post-operative markers of platelet activation (TAT, F1.2), fibrinolysis (d-dimer) and inflammation (CRP)
Use of recombinant factor VIIa after surgery to control post-operative bleeding | 48 hrs post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brian W McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada